CLINICAL TRIAL: NCT02431663
Title: Efficacy of Ketamine in Refractory Convulsive Status Epilepticus in Children: a Multicenter, Randomized, Controlled, Open-label, No-profit, With Sequential Design Study.
Brief Title: Ketamine in Refractory Convulsive Status Epilepticus
Acronym: KETASER01
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: Ospedali Riuniti Ancona (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University of Padova (Other); Bambino Gesù Hospital and Research Institute (Other); Catholic University of the Sacred Heart (Other); IRCCS Burlo Garofolo (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Nuovo Regina Margherita Hospital (Other); Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Anna Rosati, MD, PhD, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number: 2013-004396-12
Record Dates: First submitted 2015-04-03; First posted 2015-05-01 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Status Epilepticus
Keywords: refractory convulsive status epilepticus; ketamine; conventional anesthetics; children
MeSH Terms: conditions — Status Epilepticus | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketamine up to 100 mcg/kg/min (Experimental): Two intravenous boluses of 2-3 mg/kg each of ketamine will be administered 5 minutes apart and immediately followed by a continuous infusion of 5-10 mcg/kg/min. Based on both clinical or electrographic responses, dosage will be increased every 10 minutes or longer, using 2 to 10 mcg/kg/ min increments, up to 60 mcg/kg/min. Maximum duration of infusion will be of 7 days.
  Interventions: Drug: Ketamine
- midazolam & thiopental & propofol (Active Comparator): Midazolam intravenous will be increased every 5 minutes, using 2 mcg/kg/min increments, up to 12 mcg/kg/min and Thiopental intravenous will be increased every 30 minutes or longer, using 1 mg/kg/h increments, up to 6 mg/kg/h and Propofol intravenous will be increased every 5 minutes or longer, using 1 mg/kg/h increments, up to 5 mg/kg/h.
  Maximum duration of infusion for each drug will be 48 hours.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Intravenous administration in continuous
  Other Names: KETAMINA MOLTENI, vials of 2 ml (50 mg/ml)

SUMMARY:
To evaluate the efficacy of intravenous administration of ketamine in the treatment of refractory convulsive status epilepticus in children compared to administration of midazolam at high doses, thiopental and / or propofol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis and clinical EEGrafica of refractory convulsive status epilepticus
* Refractoriness of the drug I and II line
* Written informed consent from parents or legal guardian.
* Administration of rating scales in the risk of mortality (PIM III) and severity of SE (stess, status epilepticusseverity score) to be performed prior to randomization.

Exclusion Criteria:

* contraindications to the use of the medication/s in the study.
* pregnant or suspected pregnant.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2015-04; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with resolution of refractory convulsive status epilepticus | participant wil be followed for 24 hours after discontinuation of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rosati, MD, PhD, Study Chair — Children's Hospital A. Meyer of Firenze, Italy
Locations (1):
- Anna Rosati, Florence, Italy

REFERENCES:
- [Derived] Rosati A, De Masi S, Guerrini R. Ketamine for Refractory Status Epilepticus: A Systematic Review. CNS Drugs. 2018 Nov;32(11):997-1009. doi: 10.1007/s40263-018-0569-6. PMID 30232735
- [Derived] Rosati A, Ilvento L, L'Erario M, De Masi S, Biggeri A, Fabbro G, Bianchi R, Stoppa F, Fusco L, Pulitano S, Battaglia D, Pettenazzo A, Sartori S, Biban P, Fontana E, Cesaroni E, Mora D, Costa P, Meleleo R, Vittorini R, Conio A, Wolfler A, Mastrangelo M, Mondardini MC, Franzoni E, McGreevy KS, Di Simone L, Pugi A, Mirabile L, Vigevano F, Guerrini R. Efficacy of ketamine in refractory convulsive status epilepticus in children: a protocol for a sequential design, multicentre, randomised, controlled, open-label, non-profit trial (KETASER01). BMJ Open. 2016 Jun 15;6(6):e011565. doi: 10.1136/bmjopen-2016-011565. PMID 27311915